CLINICAL TRIAL: NCT00951821
Title: Concurrent Treatment for Parents and Adolescents Who Attempt Suicide
Brief Title: Concurrent Treatment for Depressed Parents and DepressedAdolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH082211 (NIH); R34MH082211 (NIH); DSIR 84 CTS; NCT00951821 (Registry Identifier: Clinical Trials.Gov)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Results first posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-03

CONDITIONS: Depression; Suicide
Keywords: Suicidal Ideation; Suicide Attempts
MeSH Terms: conditions — Depression; Suicide; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent treatment (Experimental): Concurrent treatment - experimental condition: Adolescent participants and their parents will receive concurrent cognitive behavioral therapy.
  Interventions: Behavioral: Concurrent treatment
- Adolescent treatment only (Active Comparator): Adolescent treatment only - Active Comparator: Only adolescent participants will receive cognitive behavioral therapy.
  Interventions: Behavioral: Adolescent treatment only

INTERVENTIONS:
Behavioral: Concurrent treatment — Individual CBT sessions for parents and adolescents plus combined parent-adolescent family sessions, delivered weekly for 3 months in the acute phase and bimonthly for 3 months in the maintenance phase. The techniques used to teach cognitive restructuring and problem solving to parents will be similar to those taught to the adolescents, except emotion regulation skills will be added to the parent treatment.
  Other Names: CBT for adolescents and parents
  Arms: Concurrent treatment
Behavioral: Adolescent treatment only — Individual CBT for adolescents only plus combined parent-adolescent family sessions, delivered weekly for 3 months in the acute phase and bimonthly for 3 months in the maintenance phase
  Arms: Adolescent treatment only

SUMMARY:
This study will develop an integrated treatment for adolescents who are depressed and suicidal and their parents who are depressed and have a history of suicidality.

DETAILED DESCRIPTION:
Depression, like many psychiatric disorders, has a genetic component that makes it more likely that members of the same family will have the disorder. Depression in parents, particularly mothers, may put the children at greater risk for depression. When an adolescent whose parent is depressed develops depression himself or herself, treating both the parent and the adolescent may be more effective than treating only the adolescent. This study will test a depression treatment that targets depressed suicidal adolescents with a parent or primary caretaker who is also depressed and has a history of suicidality.

Participation in this study will last 6 months. Participants will be randomly assigned to receive either concurrent parent and adolescent treatment or adolescent only treatment. For those assigned to concurrent treatment, both the adolescent participants and one of their parents will receive individual cognitive behavioral therapy (CBT) counseling sessions and joint family counseling sessions. In the adolescent only treatment condition, adolescent participants will receive individual CBT sessions, but parents will not, and both will receive joint family sessions. Counseling sessions will last 1 hour and occur weekly for 3 months, and then every other week for 3 months. CBT identifies and attempts to change problematic thought patterns. All participants will receive medication consultation if necessary.

Participants will complete assessments at baseline, post-treatment, and 6 months after completing treatment. These assessments will include questionnaires and interviews about depression, suicidal thoughts, mood regulation, behavioral problems, and family. At post-treatment and the 6-month follow-up, participants will also be asked to give feedback about the counseling, medication consultation, and their satisfaction.

ELIGIBILITY:
Inclusion Criteria for Adolescents:

* Lives at home with at least one parent or guardian
* Speaks English
* Must have made a suicide attempt and be diagnosed with major depressive disorder (MDD)

Inclusion Criteria for Primary Caretakers:

* Speaks English
* Current diagnosis of MDD and a history of suicidality

Exclusion Criteria for Adolescents:

* Judged to have developmental or cognitive delays or psychotic disorders on the basis of a standard psychiatric exam
* Diagnosis of bipolar disorder or a substance dependence (people with a diagnosis of substance abuse are eligible)
* Only one adolescent per family is eligible

Exclusion Criteria for Primary Caretakers:

* Diagnosis of bipolar disorder or substance dependence
* If taking antidepressants, not on a stable dose for 3 months

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Spirito, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Concurrent Treatment: Adolescent participants and their parents will receive concurrent cognitive behavioral therapy.
  Concurrent cognitive behavioral therapy (CBT): Individual CBT sessions for parents and adolescents plus combined parent-adolescent family sessions, delivered weekly for 3 months in the acute phase and bimonthly for 3 months in the maintenance phase. The techniques used to teach cognitive restructuring and problem solving to parents will be similar to those taught to the adolescents, except emotion regulation skills will be added to the parent treatment.
- Adolescent Treatment Only: Only adolescent participants will receive cognitive behavioral therapy.
  Adolescent only cognitive behavioral therapy (CBT): Individual CBT for adolescents only plus combined parent-adolescent family sessions, delivered weekly for 3 months in the acute phase and bimonthly for 3 months in the maintenance phase
Period: Overall Study
Arm/Group | Concurrent Treatment | Adolescent Treatment Only
Started | 16 | 8
Completed | 16 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concurrent Treatment | Adolescent Treatment Only | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.69 (1.78) | 14.0 (1.69) | 14.45 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 5 | 15
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — A standard self-report form was used for adolescents to self-identify race and ethnicity
  Participants
    Hispanic or Latino | 1 | 1 | 2
    Not Hispanic or Latino | 15 | 7 | 22
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Northeast
  participants
    United States | 16 | 8 | 24
Beck Depression Inventory [Mean (Full Range); unit: units on a scale] — Higher scores indicate greater depression; full range 0 to 60.
  units on a scale | 29.32 [8 to 49] | 19.13 [14 to 30] | 24.65 [8 to 49]
Beck Suicide Ideation Scale [Mean (Full Range); unit: units on a scale] — Higher scores indicate greater suicidal ideation; full range 0 to 38
  units on a scale | 9.81 [1 to 29] | 5.75 [0 to 15] | 8.12 [0 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory - Adolescent Report, Change in Symptom Level
Description: self-report measure of depressed mood - range of scores 0 to 60; higher scores indicate worse depression. The data in this outcome refer to change from baseline to 12 month follow-up, per the adolescent self-report.
Time Frame: 12 months
Population: intent to treat
Measure: Mean (Standard Error); unit: change in BDI (-60 to 60 possible range)
Arm/Group | Concurrent Treatment | Adolescent Treatment Only
Number analyzed (Participants) | 16 | 8
change in BDI (-60 to 60 possible range) | -17.5 (2.8) | -14.1 (3.4)
Statistical Analysis 1: Comparison: Concurrent Treatment vs Adolescent Treatment Only; Test type: Superiority or Other; p = .46, Mixed Models Analysis — Effect sizes were also calculated due to small sample size; Slope = -3.3, 95% CI 2-sided [-12.1 to 5.5] — The reported statistic (-3.3) is the difference in the change from baseline to follow-up between the two treatment arms, estimated in a mixed effect regression model

2. Secondary Outcome: Beck Suicide Scale - Adolescent Response
Description: measure of suicidal ideation - scale ranges from 0 to 38 - higher scores indicate higher suicidal ideation. These data refer to adolescent respondents. The outcome is a change score so range is from -38 to 38.
Time Frame: Measured at 12 months
Population: intent to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Concurrent Treatment | Adolescent Treatment Only
Number analyzed (Participants) | 16 | 8
units on a scale | -1.7 (1.4) | -2.1 (1.3)
Statistical Analysis 1: Comparison: Concurrent Treatment; Test type: Superiority or Other; p = .75, Mixed Models Analysis; Slope = 0.4, 95% CI 2-sided [-2.36 to 3.06] — The statistic provided (0.4) is the difference in the change in BDI score from baseline to follow-up by treatment group

ADVERSE EVENTS:
Time Frame: I year
Arm/Group | Concurrent Treatment | Adolescent Treatment Only
Serious Adverse Events (participants affected / at risk) | 5/16 | 2/8
Other Adverse Events (participants affected / at risk) | 2/16 | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Treatment (N=16) | Adolescent Treatment Only (N=8)
Inpatient Hospitalization; ED visit (Psychiatric disorders) | 5 (7) | 2 (2) — Evaluated or admitted secondary to suicidal ideation and/or behavior
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent Treatment (N=16) | Adolescent Treatment Only (N=8)
Behavior problems involving legal authorities (Psychiatric disorders) | 2 (2) | 1 (1) — Fire setting; vanda,ism

LIMITATIONS AND CAVEATS:
The outcome data from this study must be considered within the context of its limitations including the small sample size which reduces both the power to detect differences between groups as well as the stability of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No